CLINICAL TRIAL: NCT02691156
Title: Bilirubin Binding Capacity to Assess Bilirubin Load in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Smith-Kettlewell Eye Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-31187
Record Dates: First submitted 2016-02-16; First posted 2016-02-25 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Bilirubin-induced Neurologic Dysfunction; Hyperbilirubinemia; Kernicterus; Infant, Premature; Infant, Low Birth Weight
Keywords: Hematofluorometer
MeSH Terms: conditions — Hyperbilirubinemia; Kernicterus; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Premature Infants: Premature infants GA 24 to ≤34 wks at risk for hyperbilirubinemia will have BBC, ETCOc, and COHbc measured during 0-7 days of life.
  Interventions: Diagnostic Test: Bilirubin Binding Capacity; Diagnostic Test: End-tidal Carbon Monoxide; Diagnostic Test: Carboxyhemoglobin

INTERVENTIONS:
Diagnostic Test: Bilirubin Binding Capacity — Research laboratory assay of bilirubin binding capacity
  Other Names: BBC
Diagnostic Test: End-tidal Carbon Monoxide — Noninvasive bedside test to measure exhaled end-tidal carbon monoxide levels for the detection of hemolysis
  Other Names: ETCOc
Diagnostic Test: Carboxyhemoglobin — Laboratory assay of carboxyhemoglobin levels for the detection of hemolysis
  Other Names: COHbc

SUMMARY:
Most preterm newborns are managed by phototherapy to reverse hyperbilirubinemia with the intent to prevent bilirubin neurotoxicity. A threshold-based relationship between a specific total bilirubin level and need for intervention has been elusive. This is most likely due to other biomarkers such as hemolysis, developmental maturation, concurrent illnesses, or even interventions, may impede bilirubin/albumin binding. The over-prescription of phototherapy has impacted clinical and family-centered care, and in the extreme preterm infants, it may have augmented their risk of mortality. Thus, the opportunity to individualize phototherapy in in order to reduce its use is unique. The investigators have assembled a transdisciplinary team to examine critical unanswered questions including the role of bilirubin binding capacity (BBC) of an individual during the first week of life in the context of clinical modifiers and antecedents for a domain of bilirubin-induced neurologic disorders, that includes neuro-anatomical, hearing, visual and developmental processing impairments. In this study, the investigator will evaluate two new innovative nanotechniques to quantify bilirubin load for the first time in the context of a clinical decision algorithm to identify those most at risk for any bilirubin-related neurotoxicity. The investigators anticipate that knowledge gained from this study will lead to ethically testable hypotheses to individualize the prescription of phototherapy.

DETAILED DESCRIPTION:
The investigator intends to first collect simultaneous and comprehensive "acute phase" measurements of TB, BBC, ETCOc, and COHbc in MPT infants. The investigator will then seek to understand precisely the relationship between GA, TB, BBC, ETCOc, and COHbc levels and the domains of BIND. Third, The investigator will provide a comprehensive database that can be used to improve current neonatal BIND screening practices in the context of lowered and higher BBC. The investigator's working hypothesis is that exposures to modest TB levels in the presence of significantly diminished BBC in the developing neonate result in residual deficits of one or more neuroprocessing function (BIND) at TEA.

1. Patients (GA 24 to <34 wks) will be enrolled. Subject exclusion criteria: Major life-threatening anomalies and diagnosed inborn errors of metabolic disorders; attending physician or parent refusal.

   Clinical data collection: After receiving written informed consent, the research team will complete clinical data forms for infant demographics. The data forms will be consistent with and abstracted from the medical record. No additional information will be collected for this exploratory study.

   Population: The entire cohort will compromise 60-80 patients. From this cohort, 12 at-risk infants with most impaired BBC and matched with those designated as low-risk will be re-recruited for the follow-up to identify any evidence of BIND in any or all 4 of the outcome variables.

   Laboratory data: Once inclusion criteria are met, routine neonatal laboratory tests will be as clinically ordered. Each infant will tested for BBC and ETCOc at least 2 intervals (maximum 4 over 12h-7d) during rates-of-rise and -decrease in TB. Subsequent laboratory and clinical data will be paired with research data for statistical analysis.

   The investigators will compare BIND outcomes at TEA to 3 mos-corrected age (<54 wks PMA) using a re-consented sample size: n=12 for those at high risk with decreased BBC versus a GA-matched controls at low risk (n=12).
2. Measurements: 0.1-mL whole blood will be drawn in special heparinized tubes for COHbc determinations and anticoagulated blood set aside for the hematofluorometry.

Plasma for peroxidase UB assays will be stored and labeled without patient identifiers.

Frozen research samples will be transported to the Spectrum Child Health Research (SCHR) Lab for analyses. 1. BBC, TB, and UB will be measured directly: 1a. BBC, TB and UB in 50-μL whole blood using POC hematofluorometry; TB performed by the hospital-based clinical laboratory; and UB in plasma using the peroxidase method (Arrows device).

ETCOc will be determined for those breathing spontaneously.

c. Testing and techniques for outcome variables for select at-risk and matched control infants:

1. Screening ABR: Two or more simultaneously channels will consist of the electrode pairs of: 1) contralateral to ipsilateral mastoid prominence; 2) vertex to ipsilateral mastoid; and 3) vertex to contralateral mastoid for better identification of waves. Insert tubephone earphone will be used to introduce an acoustic delay to distinguish CM response from artifact. Rarefaction clicks at 90, (75), 60, (45), and 30 dBnHL will be delivered monaurally to the right and left ears. RE and LE, ≥2 repetitions, ≥2,000 sweeps/repetition. Separate recording to rarefaction and condensation clicks will be obtained at 90 dB. The surface electrical activity will be amplified x10,000 and filtered from 30-3,000 Hz. Latencies and peak-to-trough amplitudes of waves and CM from the outer hair cells in the inner ear of the ABRs will be scored independently by "masked" interpreters (Drs. Oghalia and Popelka).
2. Screening Visual Brainstem Responses after TEA (at 50-54 wks PMA): All infants in this subcohort will be evaluated using the sVEP technique described above.68 Electrodes are placed across the back of the visual cortex, midline and 2 cm to the left and right, with a reference lead at the occipital vertex. Thresholds and suprathreshold measurements will be compared with controls. Further, the infants in the bilirubin cohort can serve a case series with a dose response plot determined, comparing thresholds with TB levels. Bin averages for each type of vision can also be compared to the same for control infants to determine whether suprathreshold measures vary to any significant degree from controls (Fig. 3).

   Evidence from other studies of CNS damage suggests that lower signal amplitudes and thresholds correlate with CNS damage. Support for this sample size is based on practical considerations an ad hoc sample size calculation.
3. Neuroimaging of the brain will be performed by conventional MRI at TEA; this is the routine near-term neuroimaging for preterm infants in our institution. MRI is performed in unsedated infants, using a 3-Tesla platform with sequences that include Sagittal T1 FLAIR, Axial DWI, T2 FRFSE, FLAIR, GRE, and SSFSE, and Coronal SSFSE and 3D SPGR over 30 min. Drs. Barnes and Hintz, who will be masked to the acute phase biomarkers data, will interpret imaging utilizing a central reader form that includes white matter scoring according to a widely used classification system, and data regarding location, number, size, and imaging characteristics of lesions. Dr. Bhutani will correlate these data to the acute biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients (GA 24 to ≤34 wks)

Exclusion Criteria:

* Major life-threatening anomalies and diagnosed inborn errors of metabolic disorders
* Attending physician or parent refusal

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Inpatient premature infants
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Age-specific gradations of BBC values for each week of GA and in order to characterize degree of disordered BBC. | postnatal age 0-7 days
  This aim addresses the hypothesis that there are functional degrees and extents of BBC that can be objectively graded to quantify insufficient BBC. These data will define BBC ranges to guide objective, accurate thresholds that identify what levels of TB compared to the BBC is "safe". Infants with insufficient (>45% saturation) and near-normal (<25% saturation) BBC will be identified as select cohorts and then further tested for BIND at term-equivalent age.

SECONDARY OUTCOMES:
Determinants of bilirubin load (using rates of bilirubin production) on BBC | postnatal age 0-7 days
  This aim addresses the hypothesis that biochemical markers of bilirubin load, individually or collectively, related to excessive bilirubin production and insufficient BBC, define the mechanisms of bilirubin load for maturational age (both term PMA and GA). The studies are directed toward translating diverse components of bilirubin loads: serum albumin, BBC, and TB rate-of-rise and decrease. These data will integrate measurements of bilirubin load using established indices of bilirubin production that accurately characterize early signs of BIND at term equivalent age that may be associated with neuroanatomical changes, and NDI.

OTHER OUTCOMES:
Infants most at-risk for BIND prior to discharge (up to 55 weeks) for subtle or direct evidence of NDI at term equivalent age. | >=55 weeks PMA
  This aim addresses the hypothesis that acute phenotypic measures of BIND at TEA are identified most in preterm infants who have insufficient BBC. These data will detect perturbations in any or all domains of visuo-oculomotor, auditory, neuroanatomical (MRI) and neurodevelopmental functions.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K Bhutani, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile-Packard Children's Hospital at Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamola AA, Bhutani VK, Du L, Castillo Cuadrado M, Chen L, Shen Z, Wong RJ, Stevenson DK. Neonatal bilirubin binding capacity discerns risk of neurological dysfunction. Pediatr Res. 2015 Feb;77(2):334-9. doi: 10.1038/pr.2014.191. Epub 2014 Nov 24. PMID 25420178
- [Background] Practice parameter: management of hyperbilirubinemia in the healthy term newborn. American Academy of Pediatrics. Provisional Committee for Quality Improvement and Subcommittee on Hyperbilirubinemia. Pediatrics. 1994 Oct;94(4 Pt 1):558-65. No abstract available. PMID 7755691
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951
- [Background] Bhutani VK, Johnson LH, Shapiro SM. Kernicterus in sick and preterm infants (1999-2002): a need for an effective preventive approach. Semin Perinatol. 2004 Oct;28(5):319-25. doi: 10.1053/j.semperi.2004.09.006. PMID 15686262
- [Background] Bhutani VK, Vilms RJ, Hamerman-Johnson L. Universal bilirubin screening for severe neonatal hyperbilirubinemia. J Perinatol. 2010 Oct;30 Suppl:S6-15. doi: 10.1038/jp.2010.98. PMID 20877410
- [Background] Dennery PA, Seidman DS, Stevenson DK. Neonatal hyperbilirubinemia. N Engl J Med. 2001 Feb 22;344(8):581-90. doi: 10.1056/NEJM200102223440807. No abstract available. PMID 11207355
- [Background] Johnson L, Bhutani VK, Karp K, Sivieri EM, Shapiro SM. Clinical report from the pilot USA Kernicterus Registry (1992 to 2004). J Perinatol. 2009 Feb;29 Suppl 1:S25-45. doi: 10.1038/jp.2008.211. PMID 19177057
- [Background] Maisels MJ. What's in a name? Physiologic and pathologic jaundice: the conundrum of defining normal bilirubin levels in the newborn. Pediatrics. 2006 Aug;118(2):805-7. doi: 10.1542/peds.2006-0675. No abstract available. PMID 16882840
- [Background] Watchko JF, Maisels MJ. Jaundice in low birthweight infants: pathobiology and outcome. Arch Dis Child Fetal Neonatal Ed. 2003 Nov;88(6):F455-8. doi: 10.1136/fn.88.6.f455. PMID 14602689
- [Background] Watchko JF, Oski FA. Kernicterus in preterm newborns: past, present, and future. Pediatrics. 1992 Nov;90(5):707-15. PMID 1408544
- [Background] Morris BH, Oh W, Tyson JE, Stevenson DK, Phelps DL, O'Shea TM, McDavid GE, Perritt RL, Van Meurs KP, Vohr BR, Grisby C, Yao Q, Pedroza C, Das A, Poole WK, Carlo WA, Duara S, Laptook AR, Salhab WA, Shankaran S, Poindexter BB, Fanaroff AA, Walsh MC, Rasmussen MR, Stoll BJ, Cotten CM, Donovan EF, Ehrenkranz RA, Guillet R, Higgins RD; NICHD Neonatal Research Network. Aggressive vs. conservative phototherapy for infants with extremely low birth weight. N Engl J Med. 2008 Oct 30;359(18):1885-96. doi: 10.1056/NEJMoa0803024. PMID 18971491
- [Background] O'Shea TM, Dillard RG, Klinepeter KL, Goldstein DJ. Serum bilirubin levels, intracranial hemorrhage, and the risk of developmental problems in very low birth weight neonates. Pediatrics. 1992 Dec;90(6):888-92. PMID 1279513
- [Background] Oh W, Tyson JE, Fanaroff AA, Vohr BR, Perritt R, Stoll BJ, Ehrenkranz RA, Carlo WA, Shankaran S, Poole K, Wright LL; National Institute of Child Health and Human Development Neonatal Research Network. Association between peak serum bilirubin and neurodevelopmental outcomes in extremely low birth weight infants. Pediatrics. 2003 Oct;112(4):773-9. doi: 10.1542/peds.112.4.773. PMID 14523165
- [Background] Yeo KL, Perlman M, Hao Y, Mullaney P. Outcomes of extremely premature infants related to their peak serum bilirubin concentrations and exposure to phototherapy. Pediatrics. 1998 Dec;102(6):1426-31. doi: 10.1542/peds.102.6.1426. PMID 9832580
- [Background] Johnson L, Bhutani VK. The clinical syndrome of bilirubin-induced neurologic dysfunction. Semin Perinatol. 2011 Jun;35(3):101-13. doi: 10.1053/j.semperi.2011.02.003. PMID 21641482
- [Background] Scheidt PC, Graubard BI, Nelson KB, Hirtz DG, Hoffman HJ, Gartner LM, Bryla DA. Intelligence at six years in relation to neonatal bilirubin levels: follow-up of the National Institute of Child Health and Human Development Clinical Trial of Phototherapy. Pediatrics. 1991 Jun;87(6):797-805. PMID 2034482
- [Background] Oh W, Stevenson DK, Tyson JE, Morris BH, Ahlfors CE, Bender GJ, Wong RJ, Perritt R, Vohr BR, Van Meurs KP, Vreman HJ, Das A, Phelps DL, O'Shea TM, Higgins RD; NICHD Neonatal Research Network Bethesda MD. Influence of clinical status on the association between plasma total and unbound bilirubin and death or adverse neurodevelopmental outcomes in extremely low birth weight infants. Acta Paediatr. 2010 May;99(5):673-678. doi: 10.1111/j.1651-2227.2010.01688.x. Epub 2010 Jan 25. PMID 20105142
- [Background] Amin SB, Lamola AA. Newborn jaundice technologies: unbound bilirubin and bilirubin binding capacity in neonates. Semin Perinatol. 2011 Jun;35(3):134-40. doi: 10.1053/j.semperi.2011.02.007. PMID 21641486
- [Background] Cashore WJ, Oh W, Blumberg WE, Eisinger J, Lamola AA. Rapid fluorometric assay of bilirubin and bilirubin binding capacity in blood of jaundiced neonates: comparisons with other methods. Pediatrics. 1980 Sep;66(3):411-6. PMID 7422430
- [Background] Lamola AA, Eisinger J, Blumberg WE, Patel SC, Flores J. Flurorometric study of the partition of bilirubin among blood components: basis for rapid microassays of bilirubin and bilirubin binding capacity in whole blood. Anal Biochem. 1979 Nov 15;100(1):25-42. doi: 10.1016/0003-2697(79)90105-2. No abstract available. PMID 543536
- [Background] Hintz SR, Stevenson DK, Yao Q, Wong RJ, Das A, Van Meurs KP, Morris BH, Tyson JE, Oh W, Poole WK, Phelps DL, McDavid GE, Grisby C, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Is phototherapy exposure associated with better or worse outcomes in 501- to 1000-g-birth-weight infants? Acta Paediatr. 2011 Jul;100(7):960-5. doi: 10.1111/j.1651-2227.2011.02175.x. Epub 2011 Feb 25. PMID 21272067
- [Background] Tyson JE, Pedroza C, Langer J, Green C, Morris B, Stevenson D, Van Meurs KP, Oh W, Phelps D, O'Shea M, McDavid GE, Grisby C, Higgins R; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Does aggressive phototherapy increase mortality while decreasing profound impairment among the smallest and sickest newborns? J Perinatol. 2012 Sep;32(9):677-84. doi: 10.1038/jp.2012.64. Epub 2012 May 31. PMID 22652561
- [Background] Berlin CI, Hood LJ, Morlet T, Wilensky D, Li L, Mattingly KR, Taylor-Jeanfreau J, Keats BJ, John PS, Montgomery E, Shallop JK, Russell BA, Frisch SA. Multi-site diagnosis and management of 260 patients with auditory neuropathy/dys-synchrony (auditory neuropathy spectrum disorder). Int J Audiol. 2010 Jan;49(1):30-43. doi: 10.3109/14992020903160892. PMID 20053155
- [Background] Ahlfors CE, Wennberg RP, Ostrow JD, Tiribelli C. Unbound (free) bilirubin: improving the paradigm for evaluating neonatal jaundice. Clin Chem. 2009 Jul;55(7):1288-99. doi: 10.1373/clinchem.2008.121269. Epub 2009 May 7. PMID 19423734
- [Background] Funato M, Tamai H, Shimada S, Nakamura H. Vigintiphobia, unbound bilirubin, and auditory brainstem responses. Pediatrics. 1994 Jan;93(1):50-3. PMID 8265323
- [Background] Amin SB, Ahlfors C, Orlando MS, Dalzell LE, Merle KS, Guillet R. Bilirubin and serial auditory brainstem responses in premature infants. Pediatrics. 2001 Apr;107(4):664-70. doi: 10.1542/peds.107.4.664. PMID 11335741